CLINICAL TRIAL: NCT00326079
Title: A Study of the Glaukos Trabecular Micro-bypass Stent in Open Angle Glaucoma Subjects 1 Stent Versus 2 Stents
Brief Title: A Study of the Glaukos Trabecular Micro-bypass Stent in Open Angle Glaucoma Subjects 1 Stent Versus 2
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCF-005
Record Dates: First submitted 2006-05-12; First posted 2006-05-16 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Open-Angle Glaucoma
Keywords: Open angle; Glaucoma; Surgery
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma | interventions — Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Device: Stent
- 2 (Active Comparator)
  Interventions: Device: Stent

INTERVENTIONS:
Device: Stent — implantation of 1 Glaukos iStent versus 2 Glaukos iStents
  Other Names: iStent

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the iStent trabecular micro-bypass stent in reducing intraocular pressure (IOP) in subjects with open-angle glaucoma.

DETAILED DESCRIPTION:
The study compares 1 stent versus 2 stents.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with open-angle glaucoma (OAG)
* Subject on at least one glaucoma medication
* Signed informed consent

Exclusion Criteria:

* Angle closure glaucoma
* Secondary glaucomas except pseudoexfoliative and pigmentary; no neovascular, uveitic or angle recession glaucoma
* Prior glaucoma procedures (eg trabeculectomy, viscocanalostomy, ALT, SLT, shunt implant, collagen implant, cyclo destructive procedures etc)
* Fellow eye already enrolled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2004-08; Primary Completion 2013-05 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Efficacy | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Head of Clinical Affairs, Study Director — Glaukos Corporation
Locations (7):
- Vienna Medical University, Vienna, Austria
- Germany (3):
  - Klinik Vincentinum, Augsburg
  - Mainz University, Mainz
  - Private Practice, Weinheim
- Spain (2):
  - Hospital Clínico San Carlos, Madrid
  - Instituto Oftalmológico de Aragón, Zaragoza
- Beyoglu Eye Research and Education Hospital, Istanbul, Turkey (Türkiye)